CLINICAL TRIAL: NCT01688960
Title: A Phase 1b Study of Combined Angiogenesis Inhibition by Administering REGN910 and Aflibercept (Ziv-aflibercept) in Patients With Advanced Solid Malignancies
Brief Title: Nesvacumab (REGN910/ SAR307746) and Aflibercept ("Ziv-aflibercept" in the U.S.) in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R910-ST-1114
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Drug: nesvacumab (REGN910/ SAR307746); Drug: aflibercept (ziv-aflibercept)
- Cohort 2 (Experimental)
  Interventions: Drug: nesvacumab (REGN910/ SAR307746); Drug: aflibercept (ziv-aflibercept)
- Cohort 3a (Experimental)
  Interventions: Drug: nesvacumab (REGN910/ SAR307746); Drug: aflibercept (ziv-aflibercept)
- Cohort 3b (Experimental)
  Interventions: Drug: nesvacumab (REGN910/ SAR307746); Drug: aflibercept (ziv-aflibercept)
- Cohort 4 (Experimental)
  Interventions: Drug: nesvacumab (REGN910/ SAR307746); Drug: aflibercept (ziv-aflibercept)

INTERVENTIONS:
Drug: nesvacumab (REGN910/ SAR307746) — Dose level 1
  Arms: Cohort 1
Drug: nesvacumab (REGN910/ SAR307746) — Dose level 2
  Arms: Cohort 2; Cohort 3b
Drug: nesvacumab (REGN910/ SAR307746) — Dose level 3
  Arms: Cohort 3a; Cohort 4
Drug: aflibercept (ziv-aflibercept) — Dose level 1
  Other Names: In US: aflibercept is known as ziv-aflibercept
  Arms: Cohort 1; Cohort 2; Cohort 3a
Drug: aflibercept (ziv-aflibercept) — Dose level 2
  Other Names: In US: aflibercept is known as ziv-aflibercept
  Arms: Cohort 3b; Cohort 4

SUMMARY:
This is an open-label, multicenter, ascending, multiple dose study of nesvacumab (REGN910/ SAR307746) in combination with aflibercept ("ziv-aflibercept" in the U.S.)

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to, the following:

1. Confirmed diagnosis of solid tumor malignancy
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
3. Adequate hepatic, renal and bone marrow function
4. Resolution of toxicity from prior therapy (except alopecia) to grade less than or equal to 1

Exclusion Criteria:

Exclusion criteria include, but are not limited to, the following:

1. Patients with brain metastases, spinal cord compression, carcinomatous meningitis, or other evidence of central nervous system involvement
2. Either systolic BP greater than 140 mm Hg or diastolic BP greater than 90 mm Hg
3. Patients with medical history of myocardial infarction, unstable angina pectoris, coronary/ peripheral artery bypass graft, congestive heart failure or ventricular arrhythmia
4. Patients with deep vein thrombosis or pulmonary embolism within last 3 months
5. Patients with serious non healing wound or acute ulcer
6. Patients with treatment resistant or bleeding peptic ulcer disease, erosive esophagitis or gastritis, grade 3 or gastrointestinal bleeding/hemorrhage, infectious or inflammatory bowel disease, diverticulitis, or other uncontrolled thromboembolic event within last 3 months
7. Patients with history of abdominal or tracheal-esophageal fistula
8. Prior treatment with aflibercept (ziv-aflibercept), Ang2 or Tie2 inhibitors
9. Prior treatment with bevacizumab within last 6 weeks
10. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerable Dose (MTD) or Recommended Phase 2 Dose (RP2D) | Day 1 to Day 28
  Determine the maximum tolerable dose or recommended phase 2 dose of nesvacumab (REGN910/ SAR307746) administered in combination with aflibercept (ziv-aflibercept) in patients with advanced solid malignancies

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Day 1 to Day 170
  To assess PK parameters such as concentration of nesvacumab (REGN910/ SAR307746) and aflibercept (ziv-aflibercept).
Immunogenicity | Day 1 to Day 170
  To assess the anti-drug antibodies of nesvacumab (REGN910/ SAR307746) and aflibercept (ziv-aflibercept)
Antitumor activity | Day 1 to Day 170
  Objective tumor response according to RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1
Pharmacodynamics (PD) | Day 1 to Day 170
  Target inhibition biomarker changes, serum tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (6):
- United States (5):
  - Indianapolis, Indiana
  - New York, New York
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
- Toronto, Canada